CLINICAL TRIAL: NCT05770011
Title: Accuracy of Impression Techniques and Their Effect on the Passive Fit of Screw- Retained Bar Splinting Two Interforaminal Implants
Brief Title: Digital Versus Conventional Impression Technique in Mandibular Arch
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Bassant Sherif Gamal eldin, assistant lecturer of OMF prosthodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2351992
Record Dates: First submitted 2023-02-16; First posted 2023-03-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: one control group and two comparator groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional impression (Active Comparator): Impression will be taken conventionally using rubber base open tray
  Interventions: Device: impression material
- digital impression without splinting the scan bodies (Experimental): Impression will be taken by intraoral scaner
  Interventions: Device: intraoral scanner of nonsplinted scan bodies
- digital impression with splinting the scan bodies (Experimental): Impression will be taken by intraoral scaner
  Interventions: Device: intraoral scanner of splinted scan bodies

INTERVENTIONS:
Device: intraoral scanner of nonsplinted scan bodies — scanning of non splinted scan bodies
  Arms: digital impression without splinting the scan bodies
Device: impression material — conventional recording
  Arms: Conventional impression
Device: intraoral scanner of splinted scan bodies — scanning of splinted scan bodies
  Arms: digital impression with splinting the scan bodies

SUMMARY:
Objectives: Passive fit of screw retained frameworks is essential to avoid biological and mechanical failures in addition to transmission of unfavourable stresses to the bone-implant interface. However, Several factors contribute to the passive fit of screw retained prosthesis such as relative parallelism between the implants, implant number, impression material, impression technique and method of prothesis fabrication. The current study aims to evaluate the accuracy of three different impression techniques on the fit of screw retained bar splinting two inter-foraminal implants.

Methods: The study presents evaluation of the passive fit of screw retained bar fabricated with three different impression techniques.

DETAILED DESCRIPTION:
Surgical guide will be designed for completely edentulous patients. It will be inserted into the patient's mouth, stabilized against the upper denture and secured in place. dental implants will then be placed.

For bar fabrication using the first impression technique, closed-top primary impressions will be made followed by open top secondary impression. Extraoral scanning of the impression will be done followed by digital fabrication of the bar.

For bar fabrication using the second impression technique, scanning of the lower arch will be done using Omnicam intraoral scanner. Scanning will be done by a single calibrated operator who is trained on intraoral scanning techniques.

Scan bodies will be then screwed to the implants and scanning will be done. Both scans will be previewed on the computer desktop and superimposed together. A Standard tessellation language file will be then exported, downloaded and previewed in Inlab Exocad software .Implant system and the bar design will be selected from the software library. Then, the Standard tessellation Language file will be exported to the milling machine and milling of Cobalt chromium bar will be done.

For bar fabrication using the third technique, splinting of scan bodies will be done followed by intraoral scanning of the lower arch.

ELIGIBILITY:
Inclusion Criteria:

* - Patients' age range from 50 to 65 years old.
* Good oral hygiene is mandatory.
* Sufficient restorative space (15mm) to accept implant supported over denture diagnosed by mounting the diagnostic casts.
* Firm and healthy mucosa covering the alveolar ridge.
* Minimum bone width 5.5 mm buccolingually and of 12 mm bone height as diagnosed from the pre-operative cone beam computed tomography scan.

Exclusion Criteria:

* Heavy smokers.
* Patients with para functional habits.
* Tempromandibular Joint Disorders. (TMJ disorders)
* Patients with systemic disorders that may affect the results of this study.
* V-shaped dental arch.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
linear accuracy of impressions by superimposition | 1 year
  accurate details recorded by superimposition of the impressions using geomagic software program by measuring linear deviation in millimeters
Angular accuracy of impressions by superimposition | 1 year
  accurate details recorded by superimposition of the impressions using geomagic software program by measuring angular displacements in degrees
passive fit of screw retained bars | one year
  frame work fitting passively using screw resistance test using screw resistance parameter calculated by subtraction of passive and non passive situations angles of rotation in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Marwa El Kassaby, PhD, Study Director — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No